CLINICAL TRIAL: NCT00946972
Title: Multiple Dose Study in T2DM
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of JNJ-38431055 in Volunteers With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No safety signals were noted. The study completed the main phase, additional potential study cohorts not required.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR016447
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: JNJ-38431055; Placebo

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (explores what the body does to the drug), and pharmacodynamics (explores what a drug does to the body) of multiple doses of JNJ-38431055 in volunteers with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a double-blind (neither physician or participant knows the name of the assigned study drug), placebo-controlled (substance containing no medication), study in male and female volunteers with type 2 diabetes mellitus. For each volunteer, the study consists of a screening phase (up to 45 days), a run-in phase during which volunteers discontinue their oral anti-hyperglycemic drugs (21 to 35 days), a treatment phase during which volunteers will continue to be off their anti-hyperglycemic drugs and receive daily study drug (JNJ-38431055 or placebo) for 14 days, and a follow-up phase (10 days). After the follow-up phase, volunteers will restart their oral anti-hyperglycemic drugs. The following safety evaluations will be taken throughout the study: Electrocardiogram (an ECG is a painless procedure that gives a picture of the electrical activity of the heart), blood pressure, heart rate, and blood samples for laboratory tests. The primary outcomes will be safety and tolerability of JNJ-38431055 and 24-hour weighted mean glucose concentrations after 14 days of dosing with JNJ-38431055. Study drug will be administered as daily doses for 14 days. The two treatments will be JNJ-38431055 and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or postmenopausal or surgically sterilized females, who have type 2 diabetes mellitus
* Medically stable on the basis of physical examination, medical history, laboratory safety test results, vital signs and ECG performed at screening
* Body Mass Index (BMI) between 22 and 39.9 kg/m2, inclusive
* On a generally stable antihyperglycemic agent regimen (i.e. with no change in medication, or only 1 dose step change in dose) for at least 2 months prior to Screening visit, including volunteers who are: (a) Not currently on antihyperglycemic therapy and have an HbA1c >=7.0 % and <=10%, or (b) On a single oral antihyperglycemic agent [metformin, a sunfonylurea, a meglitinide (e.g., repaglininide or nateglinide), a DPP-IV inhibitor (sitagliptin or vildagliptin), or an alpha-glucosidase inhibitor (e.g., acarbose)] and have an HbA1c >=6.5% and <=9.5%, or (c) On low-dose dual oral agent therapy (i.e., <50% maximum labeled doses of both agents) and have an HbA1c >=6.5% and <=9.5%
* On Day -2 (two days prior to study drug administration), FPG concentrations between 120 mg/dL and 260 mg/dL, inclusive

Exclusion Criteria:

* Taking non-oral antihyperglycemic agent (e.g., insulin, exenatide or other GLP-1 analogues), or taking a thiazolidinedione (i.e., a PPARg agonist) within 3 months of the Screening visit
* History of a recent severe hypoglycemic episode, recurrent hypoglycemic episodes (i.e., within the past year), or a history of hypoglycemic unawareness
* History of clinically significant diabetic complications, including retinopathy, nephropathy, neuropathy or gastroparesis
* Positive test for alcohol and/or drugs of abuse
* Psychological and/or emotional problems, which would render the informed consent invalid, or limit the ability of the volunteer to comply with the study requirements
* Any condition that, in the opinion of the investigator, would compromise the well being of the volunteer or the study or prevent the volunteer from meeting or performing study requirements

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory values, vital signs, ECGs | Throughout the study

SECONDARY OUTCOMES:
24 hour weighted mean glucose | 24 hours
Fasting plasma glucose, glycosylated albumin | 14 days
Dose response | 14 days
Measures of beta-cell function | 14 days
Incretin levels | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.